CLINICAL TRIAL: NCT03167671
Title: The Effect of AposTherapy on Pain and Function in a Non Specific Low Back Pain Population. A Randomized Controlled Trial
Brief Title: The Effect of AposTherapy on Pain and Function in a Non Specific Low Back Pain
Acronym: AposBack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Apos Medical and Sports Technology Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-6701
Record Dates: First submitted 2017-03-21; First posted 2017-05-30 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Low Back Pain
Keywords: Oswestry; SF 36; Promis Pain and Function; Berg Balance
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Single blinded (evaluator), single-center, randomized controlled trial. Interventional and Control group with option for Control group to Cross over.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor is the only one masked in the study. They are independent of the randomization, trial coordination, and care providers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional Physical Therapy (Active Comparator): Up to 20 sessions of traditional physical therapy.
  Interventions: Other: Traditional Physical Therapy
- AposTherapy (Experimental): Treatment with at home AposTherapy with daily use of the shoe.
  Interventions: Device: AposTherapy

INTERVENTIONS:
Device: AposTherapy — AposTherapy® is a home-based exercise program utilizing footwear that causes exercise with normal daily activity
  Arms: AposTherapy
Other: Traditional Physical Therapy — Up to 20 sessions of traditional physical therapy
  Arms: Traditional Physical Therapy

SUMMARY:
AposTherapy is a home based exercise program utilizing footwear that causes exercise with normal activity that may significantly improve function in patients with back pain since patients with back pain have altered mechanics of motion contributing or due to the presence of the conditions. Capitalizing on the reported excellent adherence and clinical benefit of ApostTherapy in patients with significant knee and back pain, we propose to evaluate this as a conservative treatment that may supplant/supplement traditional pain medications and physical therapy in an at-risk urban inner city population.

DETAILED DESCRIPTION:
AposTherapy® is a home-based exercise program utilizing footwear that causes exercise with normal daily activity that may significantly improve function in patients with back pain in general, and specifically Axial Low Back Pain (NSLBP). Capitalizing on the reported excellent adherence and clinical benefit of Apos Therapy in patients with significant back pain, we propose to evaluate this as a conservative treatment that may supplant/supplement traditional pain medications and physical therapy in NSLBP population.

A possible potential use of AposTherapy® as a replacement for traditional physical therapy may yield a less costly, more effective therapy with better adherence. Problems with traditional therapy include poor patient adherence to both outpatient and home therapy programs, the added cost of travel (which may be more than $100 per session for ambulette or access-a-ride for eligible patients), and the lack of continuation in an ongoing exercise program[6-8], all of which can lead to relapse and need for retreatment. Additionally, access to physical therapy is limited for many patients since there are not enough available outpatient therapy services to meet the needs of all patients. Finding an alternative exercise program that will increase adherence, decrease total therapy visits, and improve patient's outcomes with decreased dependence on pain medications is a high priority from both patient care and cost management perspectives.

AposTherapy® potentially overcomes many of these issues by improving/modifying abnormal biomechanics (therefore decreasing pain), and providing an independent home-based exercise program utilizing footwear that causes exercise with normal activity by promoting perturbation. This biomechanical approach may significantly reduce pain and improve function in patients with nonspecific low back pain (NSLBP). Capitalizing on the reported excellent adherence and clinical benefit of AposTherapy® in patients with significant NSLBP, we propose to evaluate the biomechanical exercise (wearing an appropriately calibrated shoe at home for a prescribed amount of time each day) as a conservative treatment that may supplement or supplant traditional pain medications, interventional pain procedures and physical therapy in an at-risk urban inner city population with NSLBP.

ELIGIBILITY:
Inclusion Criteria:

* •Patients suffering from symptomatic axial lower back pain for at least 24 weeks.

  * Patients with VAS pain score of ≥3cm (measured at baseline).
  * Males and females between the ages of 30-85.
  * 17<BMI<40
  * Ambulatory and active patients that can participate in a rehabilitation program that includes daily walking
  * Stable medicine regimen (no recent changes to their pain medication within a month)
  * Able to walk at least 50 meters and scored positive on the STEADI test (Supp. 1)
  * Able to understand, read and sign the informed consent form
  * English or Spanish speaking

Exclusion Criteria:

* •Patients suffering from active inflammatory joint disease.

  * Patients with diagnosis of neuromuscular disease.
  * Patients with more than 3 falls in the last 52 weeks, OR any balance related fall with an injury in the last 52 weeks.
  * Patients exhibiting a lack of physical or mental ability to perform or comply with the study procedure.
  * Patients with a history of pathological osteoporotic fracture
  * Patients with referred pain consistent with radicular etiology
  * Patients with generalized body pain (both upper and lower extremities).
  * No spine surgery within 24 weeks.
  * No image guided lumbar intervention in the past 8 weeks.
  * No major cardiovascular comorbidities (able to enroll in an active exercise program)
  * Patient started on lipid lowering medication in last 12 weeks
  * Any change in blood pressure medications
  * No recent physical therapy for the back. (within the last 12 weeks)
  * No active heart disease (ischemia or heart failure admissions within 24 weeks) and no active COPD (exacerbation within 24 weeks)
  * No active malignancies on ongoing treatment
  * Patient with neurological gait pattern.
  * Patient requiring assistive device during gait analysis.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Function | 1 Year
  Improvement in back pain measured and assessed with the Oswestry Disability Index (ODI).

SECONDARY OUTCOMES:
PROMIS (Patient-Reported Outcomes Measurement Information System) Pain Interference and Physical Function | 1 year
  Pain and Function measured through PROMIS short forms
Pain medication consumption | 1 year
  medication consumption
Quality of life survey | 1 year
  Quality of life assessed with Short Form Health Survey questionnaire
Gait assessment | 1 year
  objective analysis of patients' gait assessed with a pressure mat to demonstrate stride length, velocity, and symmetry.
6-min walk test | 1 year
  objective assessment using maximum distance comfortably walked in 6 minutes on a 100 foot closed course
Dynamic balance | 1 year
  Measured by Berg balance test assessed with a questionnaire
Static balance | 1 year
  functional reach test assessed by physically testing the patient with a standardized set of instructions
Blood pressure | 1 year
  Change in blood pressure , physiological parameter
resting heart rate | 1 year
  change in resting heart rate , physiological parameter
Overall activity | 1 year
  overall activity measured as daily steps, through wristband devices
sleep patterns | 1 year
  Total sleep time measured in minutes through wristband activity monitor (FitBit) measured over one week
Visual Analog Scale (VAS) for pain measurement | 1 year
  questionnaire
Medication Consumption | 1 year
  Track increase or decrease in Medication consumption- assessed through patient interview and patent report
Medication Costs | 1 year
  Calculate monetary savings in Medication Costs- assessed through patient interview and prevailing market cost information
Hospitalization utilizations | 1 year
  Calculate the increase/decrease in hospital facility utilization - assessed with patient interview and health records.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew N Bartels, MD, MPH, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freburger JK, Holmes GM, Agans RP, Jackman AM, Darter JD, Wallace AS, Castel LD, Kalsbeek WD, Carey TS. The rising prevalence of chronic low back pain. Arch Intern Med. 2009 Feb 9;169(3):251-8. doi: 10.1001/archinternmed.2008.543. PMID 19204216
- [Background] Meucci RD, Fassa AG, Faria NM. Prevalence of chronic low back pain: systematic review. Rev Saude Publica. 2015;49:1. doi: 10.1590/S0034-8910.2015049005874. Epub 2015 Oct 20. PMID 26487293
- [Background] Woolf AD, Pfleger B. Burden of major musculoskeletal conditions. Bull World Health Organ. 2003;81(9):646-56. Epub 2003 Nov 14. PMID 14710506
- [Background] Hayden JA, van Tulder MW, Malmivaara AV, Koes BW. Meta-analysis: exercise therapy for nonspecific low back pain. Ann Intern Med. 2005 May 3;142(9):765-75. doi: 10.7326/0003-4819-142-9-200505030-00013. PMID 15867409
- [Background] Tsao H, Hodges PW. Immediate changes in feedforward postural adjustments following voluntary motor training. Exp Brain Res. 2007 Aug;181(4):537-46. doi: 10.1007/s00221-007-0950-z. Epub 2007 May 3. PMID 17476489
- [Background] Hides JA, Jull GA, Richardson CA. Long-term effects of specific stabilizing exercises for first-episode low back pain. Spine (Phila Pa 1976). 2001 Jun 1;26(11):E243-8. doi: 10.1097/00007632-200106010-00004. PMID 11389408
- [Background] Keefe FJ, Hill RW. An objective approach to quantifying pain behavior and gait patterns in low back pain patients. Pain. 1985 Feb;21(2):153-161. doi: 10.1016/0304-3959(85)90285-4. PMID 3157094
- Available data/document: Book: ISBN-10: 1886039224 — https://www.amazon.com/Prescription-Drug-Abuse-Epidemic-Understanding/dp/1886039224